CLINICAL TRIAL: NCT06241573
Title: Lunsayil LTE: An Extension Trial Assessing Long-term Spesolimab Treatment in Patients With Hidradenitis Suppurativa (HS)
Brief Title: A Study to Test Long-term Treatment With Spesolimab in People With a Skin Condition Disease Called Hidradenitis Suppurativa (HS) Who Took Part in a Previous Study With Spesolimab
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1368-0130; 2023-508377-82-00 (Registry Identifier: CTIS (EU)); U1111-1300-2310 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2024-01-29; First posted 2024-02-05 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Hidradenitis Suppurativa (HS)
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — spesolimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Patients treated in Part I of parent trial 1368-0098 (NCT05819398) (Experimental)
  Interventions: Drug: Spesolimab
- Patients treated in Part II of parent trial 1368-0098 (NCT05819398) (Experimental)
  Interventions: Drug: Spesolimab
- Patients treated in parent trial 1368-0100 (Experimental)
  Interventions: Drug: Spesolimab

INTERVENTIONS:
Drug: Spesolimab — Spesolimab

SUMMARY:
This study is open to people with hidradenitis suppurativa (HS) who have completed another study with spesolimab (study 1368-0098 (NCT05819398) or study 1368-0100).

The purpose of this study is to find out how well people tolerate spesolimab and whether it helps people with HS in the long-term. For about 1.5 years, participants get spesolimab injections under the skin every 2 weeks.

Participants are in the study for about 2 years. During this time, participants have 41 visits. 24 visits are done at the study site. 17 visits can be done by video call at the participant's home. At study visits, doctors check the severity of the participant's HS and collect information on any health problems of the participants.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated written informed consent in accordance with ICH Harmonized Guideline for Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial.
2. Participants must be within the defined Residual Effect Period corresponding to 16 weeks since last spesolimab administration.
3. Participants who have completed treatment in the parent hidradenitis suppurativa (HS) spesolimab trial (1368-0098 (NCT05819398) or 1368-0100) without premature discontinuation and are willing and able to continue treatment in this trial.
4. Woman of childbearing potential (WOCBP) must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly.

Exclusion Criteria:

1. Women who are pregnant, nursing, or who plan to become pregnant while in the trial.
2. Use of any drug considered by the investigator likely to interfere with the safe conduct of the trial since the last visit of the parent trials.
3. Use of immunomodulatory biologics or investigational agents since the last visit of the parent trials.
4. Participants who require / intend to use certain restricted medications such as immunomodulatory biologics or other investigational drugs/devices during the course of the trial.
5. Relevant chronic or acute infections including human immunodeficiency virus (HIV) and viral hepatitis. The corresponding laboratory tests will be performed at Visit 1. A participant can be re-screened if the participant was treated and is cured from the acute infection.

Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2024-05-08 (Actual); Primary Completion 2025-04-11 (Actual); Study Completion 2025-04-11 (Actual)

PRIMARY OUTCOMES:
Occurrence of treatment emergent adverse events (TEAE) | up to 92 weeks

CONTACTS AND LOCATIONS:
Locations (36):
- United States (4):
  - First OC Dermatology, Fountain Valley, California
  - Dermatology Research Associates, Los Angeles, California
  - Integrative Skin Science and Research-Sacramento-69402, Sacramento, California
  - Clinical Trials Research Institute, Thousand Oaks, California
- Argentina (3):
  - STAT Research, CABA
  - Hospital Italiano de Buenos Aires, CABA
  - Hospital Alemán, Capital Federal
- Australia (2):
  - Holdsworth House Medical Practice, Sydney, New South Wales
  - Alfred Hospital, Melbourne, Victoria
- Bulgaria (2):
  - Medical Center "Kordis", Pleven
  - ASMC-IPSMC-skin and Veneral Diseases, Sofia
- Canada (3):
  - SimcoDerm Medical and Surgical Dermatology Centre, Barrie, Ontario
  - Guelph Dermatology Research, Guelph, Ontario
  - Dr. S. K. Siddha Medicine Professional Corporation, Newmarket, Ontario
- France (2):
  - HOP Privé Antony, Antony
  - HOP Edouard Herriot, Lyon
- Germany (2):
  - Fachklinik Bad Bentheim, Bad Bentheim
  - Hautmedizin Saar, Merzig
- Japan (5):
  - Kurume University Hospital, Fukuoka, Kurume
  - Ogaki Municipal Hospital, Gifu, Ogaki
  - The University of Tokyo Hospital, Tokyo, Bunkyo-ku
  - Nihon University Itabashi Hospital, Tokyo, Itabashi-ku
  - Tokyo Medical University Hospital, Tokyo, Shinjuku-ku
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kauno Klinikos, Kaunas
  - Vilnius University Hospital, Santariskiu, Vilnius
- Malaysia (5):
  - Hospital Pulau Pinang-Pulau Pinang-21953, Georgetown Pulau Pinang
  - Hospital Sultan Ismail, Johor Bahru
  - Hospital Kuala Lumpur, Kuala Lumpur
  - Sarawak General Hospital, Kuching
  - Sunway Medical Centre, Selangor Darul Ehsan
- Poland (3):
  - Non-Public Health Care Facility LABDERM, Ossy
  - Provita Clinic, Warsaw
  - Royalderm, Warsaw
- National University Hospital-Singapore-42005, Singapore, Singapore
- Seoul National University Hospital, Seoul, South Korea
- Hospital Universitario Miguel Servet, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com